CLINICAL TRIAL: NCT03451786
Title: A Multi-center, Prospective Clinical Trial to Evaluate the Safety and Effectiveness of a Posterior Chamber Intraocular Lens for Correction of Aphakia Following Cataract Removal
Brief Title: Prospective Clinical Trial to Evaluate the Safety and Effectiveness of the IOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Estelle Poineau (Industry)
Responsible Party: Sponsor-Investigator, Estelle Poineau, Clinical Project Manager, Carl Zeiss Meditec AG
Organization: Carl Zeiss Meditec AG (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONT-301-17
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Results first posted 2022-02-01 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Cataract Unilateral; Aphakia
MeSH Terms: conditions — Aphakia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment group (Experimental)
  Interventions: Device: IOL

INTERVENTIONS:
Device: IOL — Intraocular lens

SUMMARY:
To establish the safety and effectiveness of the CT LUCIA 611P posterior chamber intraocular lens for the correction of aphakia following extracapsular cataract extraction via phacoemulsification in adult patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 22 years or older at the time of study enrollment.
2. Visually significant cataract in the study eye for which phacoemulsification cataract extraction and posterior chamber IOL implantation is indicated.
3. Projected postoperative BCDVA 0.20 logMAR or better in the study eye, as determined by Investigator's medical judgment.
4. Calculated spherical power targeted at emmetropia at distance in the study eye.
5. Calculated IOL power between +4.0 D and +34.0 D, inclusive, in the study eye.
6. If wearing rigid gas permeable (RGP) contact lens in the study eye, willingness to discontinue lens wear for ≥ 30 days prior to preoperative biometry.
7. Availability, willingness, and sufficient cognitive awareness to return for study-required visits and comply with examination procedures.
8. Willingness to sign the IRB-approved informed consent form (ICF) for study participation.

Exclusion Criteria:

1. Mature cataract in the study eye that is likely to prolong surgical procedure and/or lead to intraoperative complications prior to attempted IOL implantation.
2. Planned cataract removal using a femtosecond laser.
3. Any visually significant intraocular media opacity other than cataract in the study eye (as determined by the investigator).
4. Significant refractive error (hyperopia/myopia) of axial or pathologic origin in the study eye that, in the judgment of the investigator, could confound outcomes.
5. Abnormal corneal findings in either eye (e.g. keratoconus, pellucid marginal degeneration, or irregular astigmatism).
6. Any anterior segment pathology in the study eye that could significantly affect outcomes (e.g. chronic uveitis, iritis, aniridia, rubeosis iridis, clinically significant corneal or anterior membrane dystrophies, poor pupil dilation, etc.)
7. Any condition in the study eye that could affect IOL stability (e.g. pseudoexfoliation, zonular dialysis, evident zonular weakness or dehiscence, etc.).
8. History of severe dry eye in the study eye that, in the judgment of the investigator, would impair the ability to obtain reliable study measurements.
9. History of serious corneal disease (e.g., herpes simplex, herpes zoster keratitis, etc.) in either eye.
10. History of any clinically significant retinal pathology or ocular diagnosis (e.g. diabetic retinopathy, ischemic diseases, macular degeneration, retinal detachment, optic neuropathy, amblyopia, strabismus, microphthalmos, aniridia, epiretinal membrane etc.) in the study eye that could alter or limit final postoperative visual prognosis.
11. History of cystoid macular edema in either eye.
12. History of uveitis in either eye.
13. History of intraocular or corneal surgery in the study eye.
14. Uncontrolled glaucoma in the study eye (per Investigator judgment).
15. Current ocular infection in the study eye.
16. Fellow eye BCDVA worse than 1.0 logMAR.
17. Presence of uncontrolled systemic disease that could increase operative risk (e.g., diabetes mellitus, active cancer treatment, mental illness, dementia, immunocompromised, connective tissue disease, clinically significant atopic disease, etc.).
18. Use of or history of use of systemic medications with significant ocular side effects or any medications that could confound the outcome or increase patient risk (e.g., steroids, Tamsulosin Hydrochloride [Flomax] or other medications including anticholinergics or alpha-adrenergic blocking agents with similar side effects [e.g. small pupil/floppy iris syndrome], anti-metabolites, etc.)
19. Participation in any other non-eye related drug or device clinical trial within 30 days prior to enrolling in this study and/or during study participation.
20. Participation in any eye-related drug or device clinical trial within 90 days prior to enrolling in this study and/or during the study participation.
21. Planned concomitant ocular procedure during cataract surgery (e.g., glaucoma surgery including implantation of MIGS, astigmatic correction surgery, penetrating keratoplasty [PK], laser-assisted in situ keratomileusis [LASIK], etc.)
22. Pregnant, lactating or, if able to bear children, unwilling to use medically acceptable birth control over the course of the study.
23. Unsuitable for study participation for any other reason, as determined by Investigator's clinical judgment (reason to be documented on eCRF).

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 369 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Argus Research at Cape Coral Eye Center, Cape Coral, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schallhorn SC, Bonilla M, Pantanelli SM. Outcomes of a multicenter U.S. clinical trial of a new monofocal single-piece hydrophobic acrylic IOL. J Cataract Refract Surg. 2022 Oct 1;48(10):1126-1133. doi: 10.1097/j.jcrs.0000000000000943. Epub 2022 Mar 25. PMID 35333839

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Group
Started | 369
Completed | 310
Not Completed | 59

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Group
Number analyzed (Participants) | 339
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.1 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 208
  Male | 131
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18
  Not Hispanic or Latino | 321
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 29
  White | 299
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Best Corrected Distance Visual Acuity
Description: Proportion of subjects achieving BCDVA 0.3 logMAR or better
Time Frame: postoperative days 330-420
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 310
Participants | 308

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/339
Serious Adverse Events (participants affected / at risk) | 13/339
Other Adverse Events (participants affected / at risk) | 32/339
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=339)
Retinal detachment (Eye disorders) | 1 (1)
Anterior capsular contraction (Eye disorders) | 1 (1)
Acute myocardial infraction (Cardiac disorders) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1)
Aortic aneurysm (Cardiac disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Hip fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Post procedural complication (Surgical and medical procedures) | 1 (1)
Post procedural hemorrhage (Surgical and medical procedures) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Spinal compression fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Unevaluable event (General disorders) | 1 (1)
Chronic kidney disease (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=339)
cystoid macular edema (Eye disorders) | 7 (7)
Intraocular pressure increased (Eye disorders) | 25 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-12-21): https://cdn.clinicaltrials.gov/large-docs/86/NCT03451786/Prot_001.pdf